CLINICAL TRIAL: NCT06318572
Title: Desarrollo de Programas de intervención psicológica Autoadministrable Con Soporte de Nuevas tecnologías Como Tratamiento Para Pacientes Con Trastornos Funcionales Digestivos.
Brief Title: Development of Self-administrable Psychological Intervention Programs Supported by New Technologies as a Treatment for Patients With Functional Digestive Disorders.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)166/2021
Record Dates: First submitted 2024-02-22; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological intervention (Experimental)
  Interventions: Behavioral: Psychological intervention
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Psychological intervention — Patients will have 3 visits during the 7 weeks study length. On day -7 a first visit will be made verifying that inclusion criteria are met, the informed consent will be obtained and a rectal sensitivity test will be performed. A symptom questionnaire will be delivered to the patient for daily assessment of gastrointestinal symptoms.
  On day 0, a stool sample will be collected and the symptom questionnaire will be reviewed to confirm inclusion criteria. Patients will begin the program of psychological intervention. A first, session of psychoeducation will be performed, and thereafter sessions of psychotherapy will be performed at home during 6 weeks.
  At the end of treatment a last visit will be performed, collecting the symptoms scored during the last 7 days. A new stool sample will be collected and a rectal sensitivity study will be performed.
  Severity of symptom questionnaire will be filled at the beginning, after 3 weeks, at the end of the treatment, at 3 months and at 6 months.
  Arms: Psychological intervention
Behavioral: Placebo — Patients will have 3 visits during the 7 weeks study length. On day -7 a first visit will be made verifying that inclusion criteria are met, the informed consent will be obtained and a rectal sensitivity test will be performed. A symptom questionnaire will be delivered to the patient for daily assessment of gastrointestinal symptoms.
  On day 0, a stool sample will be collected and the symptom questionnaire will be reviewed to confirm inclusion criteria. Patients will be instructed to take a capsule containing 0.5 g during 6 weeks.
  At the end of treatment a last visit will be performed, collecting the symptoms scored during the last 7 days, A new stool sample will be collected and a rectal sensitivity study will be performed.
  Severity of symptom questionnaire will be filled at the beginning, after 3 weeks, at the end of the treatment, at 3 months and at 6 months.
  Arms: Placebo

SUMMARY:
Disorders of gut-brain interaction (DGBI) are produced by disturbances in the interplay between the gut and the central nervous system. Several psychological factors like anxiety, depression and altered coping are over-represented in these disorders. Recent surveys have shown that DGBI affect up to 40 % of the general population.

Psychological interventions like cognitive behavioral therapy and hypnosis have been shown to be beneficial for managing these disorders. However, access to psychological interventions is very limited due to lack of resources to treat these very frequent conditions.

OBJECTIVE: To determine the effects of psychological interventions using specifically developed therapeutic programs based on virtual reality, for telematic use at home, on symptoms severity, comorbidities, visceral sensitivity and intestinal dysbiosis in patients with DGBI.

METHODOLOGY: After development of a program of psycho-education on DGBI using interactive immersion by means of virtual reality (VR) a randomized clinical trial will be developed. Consecutive patients will be randomized 1:1 to active treatment or placebo. In each patient in the active treatment group a session of psychoeducation using specifically developed VR-video leaded by a gastroenterologists, will be followed by telematic weekly group sessions of psycho-education leaded by a psychologist. During the 6 weeks of the treatment period patients will be instructed to perform self-administrable sessions of psychotherapy at home (by means VR). Patients in the placebo group willl take a placebo capsule daily.

OUTCOME MEASURES. In all patients, severity of symptoms (primary outcome), QoL, somatic and psychological comorbidities (using specific questionnaires), visceral sensitivity (by means of a barostat) and microbiota analysis, will be performed before and at the end of the treatment period. Symptom severity will be assess also in follow-up phone calls at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI (Body Mass Index) between 18.5-24.99, with variations of up to 15%.
* Ability to understand instructions and follow protocol.
* Access to internet network from usual residence.

Exclusion Criteria:

* Previous history of abdominal surgery with the exception of appendectomy and herniorrhaphy.
* Abuse of alcohol, tobacco or narcotics.
* Medical evidence of organic gastrointestinal pathology, hepatopathy, endocrinopathy, heart disease or contagious disease, as well as major psychiatric disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Severity of abdominal symptoms | 6 months
  Changes from basal scores in the severity of abdominal symptoms will be calculated using the irritable bowel syndrome-symptom severity score (IBS-SSS), where score 0 is the lack of symptoms, and score 500 is maximal severity of symptoms.

SECONDARY OUTCOMES:
IBS related Quality of life | 6 weeks
  Changes from basal scores in the IBS related quality of life will be calculated using the irritable Bowel Syndrome Quality of Life Questionnaires (IBS-QoL). Rated from 0-100 % (worst-best quality of life).
Stress | 6 weeks
  Changes from basal scores in the patients perceived stress will be calculated using the perceived stress scale (PSS). Score range 0 (no stress-40 highest perceived stress).
Anxiety and depression | 6 weeks
  Changes from basal scores in the anxiety and depression rated by patients will be calculated using the hospital anxiety and depression scale (HAD). Score range 0 (no anxiety/depression-21 highest anxiety and depression in the respective scales).
Somatic co-morbidities | 6 weeks
  Changes from basal scores in the somatic co-morbidities will be calculated using the personal health questionnaire (PHQ-15). Score range 0 (no somatization-30 highest somatization).
Rectal sensitivity | 6 weeks
  Changes from basal scores in the sensitivity induced by progressive rectal distension applied by means of a barostat, will be calculated using a 0 (no perception)-6 (painful sensation) score scale.
Analysis of gut microbiota composition | 6 weeks
  Changes from basal scores in the alfa and beta diversity and relative abundance of gut microbes will be calculated using 16S rRNA bacterial metagenomic sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain